CLINICAL TRIAL: NCT05096832
Title: A Global, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Phase III Clinical Study to Evaluate the Efficacy, Safety, and Immunogenicity of Sequential Immunization of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) Against COVID-19 in Healthy Adults Aged 18 Years and Older After the Vaccination of 2 Doses of Inactivated Vaccines
Brief Title: Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) Booster Study
Acronym: COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TG2102V01
Record Dates: First submitted 2021-10-21; First posted 2021-10-27 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Pandemic
Keywords: V-01 Booster
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V-01 COVID-19 Vaccine (Experimental): 1 dose on Day 0, which should be 3-6 months after the second dose of 2-dose regimen of inactive vaccine (BBIBP-CorV or CoronaVac).
  Interventions: Biological: Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01)
- Placebo control (Placebo Comparator): 1 dose on Day 0, which should be 3-6 months after the second dose of 2-dose regimen of inactive vaccine (BBIBP-CorV or CoronaVac).
  Interventions: Biological: Blank Preparation of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01)

INTERVENTIONS:
Biological: Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) — Appearance: Creamy white suspension Dosage form: Suspension for injection Strength: 10 μg (0.5 mL) /vial Vaccination route: Intramuscular injection into the lateral deltoid of the upper arm Vaccination dosage: 10 μg (0.5 mL) Immunization schedule: 1 dose on Day 0, which should be 3-6 months after the second dose of 2-dose regimen of inactive vaccine (BBIBP-CorV or CoronaVac).
  Storage condition: Store at 2-8 °C protected from light Expiry date: 24 months temporarily
  Other Names: V-01
  Arms: V-01 COVID-19 Vaccine
Biological: Blank Preparation of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) — The dosage, appearance, administration method, and other aspects are consistent with that of investigational vaccine, except that no vaccine antigen is contained.
  Other Names: Placbo
  Arms: Placebo control

SUMMARY:
A Global, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Phase III Clinical Study to Evaluate the Efficacy, Safety, and Immunogenicity of Sequential Immunization of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) Against COVID-19 in Healthy Adults Aged 18 Years and Older after the Vaccination of 2 Doses of Inactivated Vaccines

DETAILED DESCRIPTION:
This is a global, multicenter, randomized, double-blind, placebo-controlled phase III clinical study. Approximately 10,722 participants aged 18 years and older who have completed the 2 doses of administration of inactive vaccines (BBIBP-CorV or CoronaVac) will be enrolled in this study to evaluate the efficacy, safety and immunogenicity of V-01.

The eligible participants will be randomly assigned to receive dose of either 10 μg V-01 or a placebo in a 1:1 randomization ratio. Assignment will be stratified by age (18-59 years vs. ≥ 60 years), gender (male vs. female), whether or not being enrolled into immunogenicity subgroup (yes vs no), and the types of inactivated vaccines (BBIBP-CorV vs. CoronaVac).

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Voluntarily participate in the study and sign the informed consent form.
2. Adults aged 18 years and older at time of consent, male or female.
3. Able to and willing to comply with study procedure based on the assessment of the investigator.
4. Participants who have completed the second dose of 2-dose regimen of inactive vaccination (BBIBP-CorV or CoronaVac) against SARS-CoV-2 in the past 3-6 months (Note: Participants who received mixed vaccination of BBIBP-CorV and CoronaVac will not be enrolled).
5. Healthy participants or participants with pre-existing stable medical conditions (A stable medical condition is defined as a disease not requiring significant change in therapy or hospitalization for worsening disease within 3 months before enrollment).
6. Males of reproductive potential and females of childbearing potential voluntarily agree to take effective and acceptable contraceptive methods from the signing of informed consent form to 3 months after vaccination; and a female participant of childbearing potential should have a negative pregnancy test at screening and on the day of vaccination (day 0).

Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, hysterectomy) or postmenopausal (defined as amenorrhea for ≥ 12 consecutive months prior to screening without an alternative medical cause).

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. History of previous COVID-19 infection.
2. Positive for SARS-CoV-2 test by RT-PCR during screening period (Note: Participants can be enrolled in the study and receive the investigational product without waiting for the report of the SARS-CoV-2 test by RT-PCR).
3. History of severe acute respiratory syndrome (SARS), Middle East respiratory syndrome (MERS), and other human coronavirus infections or diseases.
4. History of severe allergy to any vaccine, e.g., acute allergic reactions, urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain etc., or be allergic to any components of V-01.
5. Any confirmed or suspected immunosuppression or immunodeficiency condition known from medical history, including human immunodeficiency virus (HIV) infection, asplenia.
6. Serious or uncontrolled cardiovascular diseases, nervous system disorders (e.g., Guillain-Barre syndrome), blood and lymphatic system disorders, immune system disorders, hepatorenal disorders, respiratory system disorders (e.g., active tuberculosis, pulmonary fibrosis), metabolic and skeletal systems disorders or malignant tumors (except for skin basal cell carcinoma or in situ carcinoma of uterine cervix that has been cured for more than 5 years).
7. Hereditary hemorrhagic tendency or coagulation dysfunction, or a history of thrombosis or hemorrhagic disease, or requirement of continuous use of anticoagulants.
8. Prior use of any medication to prevent COVID-19 within 1 week before signing the informed consent form (except for previous vaccines, BBIBP-CorV or CoronaVac), e.g., use of antipyretics without pyrexia and any other symptoms.
9. Received attenuated live vaccine within 28 days before the vaccination or any other vaccines (licensed or investigational) within 14 days before the vaccination.
10. Has participated in an interventional clinical study within 1 months prior to the day of vaccination.
11. Injection of immunoglobulin and/or other blood products within 3 months before the administration of study vaccine.
12. Long-term use (continuous use > 14 days) of glucocorticoids (≥ 10 mg/day of prednisone or its equivalent dose) or other immunosuppressive agents within 6 months before signing the informed consent form; however, enrollment is allowed for the following conditions: inhaled or topical use of topical steroids, or short-term use (treatment course ≤ 14 days) of oral steroids.
13. Pregnant or breastfeeding women.
14. Planning to donate blood during the study period.
15. Suspected or known alcohol or drug dependence.
16. History of severe psychiatric disorders which may affect study participation.
17. Planning to permanently move from the local area before study completion or leave the local area for a long time during the period of study visits, so that the scheduled visits cannot be followed.
18. Those considered by the investigator as inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10381 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
the relative efficacy of recombinant SARS-CoV-2 fusion protein vaccine (V-01) as a booster to prevent symptomatic and RT-PCR positive COVID-19 (mild or above severity) | From 15days after the administration of recombinant SARS-CoV-2fusion protein vaccine (V-01) to 12 months after full-courseimmunization
  To evaluate the relative efficacy of recombinant SARS-CoV-2 fusion protein vaccine (V-01) as a booster to prevent symptomatic and reverse transcription polymerase chain reaction (RT-PCR) positive COVID-19 (mild or above severity) compared with the placebo control group.
The incidence of adverse events (AEs) | Within 28 days after the booster vaccination
  To evaluate the incidence of adverse events (AEs) within 28 days after the booster vaccination.

SECONDARY OUTCOMES:
The relative vaccine efficacy of V-01 as a booster to prevent severe or above COVID-19 | From 15days after the administration of recombinant SARS-CoV-2fusion protein vaccine (V-01) to 12 months after full-courseimmunization
  To evaluate the relative vaccine efficacy of V-01 as a booster to prevent severe or above COVID-19 compared with the placebo control group.
The relative vaccine efficacy of V-01 as a booster to prevent symptomatic and RT-PCR positive COVID-19 (mild or above severity) | From 15days after the administration of recombinant SARS-CoV-2fusion protein vaccine (V-01) to 12 months after full-courseimmunization
  To evaluate the relative vaccine efficacy of V-01 as a booster to prevent symptomatic and RT-PCR positive COVID-19 (mild or above severity) in different age subgroups compared with the placebo control group.
The relative vaccine efficacy of V-01 as a booster to prevent suspected but not confirmed COVID-19 | From 15days after the administration of recombinant SARS-CoV-2fusion protein vaccine (V-01) to 12 months after full-courseimmunization
  To evaluate the relative vaccine efficacy of V-01 as a booster to prevent suspected but not confirmed COVID-19 compared with the placebo control group.
The relative vaccine efficacy of V-01 as a booster to prevent death caused by COVID-19 | From 15days after the administration of recombinant SARS-CoV-2fusion protein vaccine (V-01) to 12 months after full-courseimmunization
  To evaluate the relative vaccine efficacy of V-01 as a booster to prevent death caused by COVID-19 compared with the placebo control group.
The relative vaccine efficacy of V-01 as a booster to prevent hospitalization caused by COVID-19 | From 15days after the administration of recombinant SARS-CoV-2fusion protein vaccine (V-01) to 12 months after full-courseimmunization
  To evaluate the relative vaccine efficacy of V-01 as a booster to prevent hospitalization caused by COVID-19 compared with the placebo control group.
The incidence of serious adverse events (SAEs) and adverse events of special interest (AESIs) | Within 12 months after the booster vaccination
  To evaluate the incidence of serious adverse events (SAEs) and adverse events of special interest (AESIs) within 12 months after the booster vaccination.
The seroconversion rate of serum SARS-CoV-2 RBD protein-binding antibody, GMT and GMI (Immunology Subgroup Only) | At day 14, day 28, month 3, month 6, and month 12 after immunization
  To evaluate the immunogenicity of V-01.

OTHER OUTCOMES:
The genotype of SARS-CoV-2 in symptomatic and RT-PCR positive COVID-19 cases. | From the administration of recombinant SARS-CoV-2fusion protein vaccine (V-01) to 12 months after immunization
  To explore the genotype of SARS-CoV-2 in symptomatic and RT-PCR positive COVID-19 cases.
Immunogenicity of V-01 against new SARS-CoV-2 variants | From the administration of recombinant SARS-CoV-2fusion protein vaccine (V-01) to 12 months after immunization
  To explore the immunogenicity of V-01 against new SARS-CoV-2 variants.

CONTACTS AND LOCATIONS:
Locations (18):
- Malaysia (10):
  - Sarawak General Hospital, Kuching, Sarawak
  - Sunway Medical Centre Velocity (SMCV) Cheras, Kuala Lumpur
  - Hospital Pakar Sultanah Fatimah, Muar town
  - Sunway Medical Centre (SunMed), Petaling Jaya
  - Hospital Pulau Pinang, Pulau Pinang
  - Klinik Kesihatan Seremban 2, Seremban
  - Seri Manjung Hospital, Seri Manjung
  - Hospital Sibu, Sibu
  - Hospital Sultan Abdul Halim, Sungai Petani
  - Hospital Taiping, Taiping
- Pakistan (8):
  - Central Hospital Gujranwala, Gujranwala
  - Shifa International Hospitals, Islamabad
  - Aga Khan University Hospital, Karachi
  - Dow University Hospital, Karachi
  - Sindh Infectious Diseases Hospital & Research Center, Karachi
  - Al Khidmat Foundation - Surraya Azeem Waqf Hospital, Lahore
  - Avicenna Dental College, Lahore
  - Central Park Medical College and Hospital, Lahore

REFERENCES:
- [Derived] Wang XY, Mahmood SF, Jin F, Cheah WK, Ahmad M, Sohail MA, Ahmad W, Suppan VK, Sayeed MA, Luxmi S, Teo AH, Lee LY, Qi YY, Pei RJ, Deng W, Xu ZH, Yang JM, Zhang Y, Guan WX, Yu X. Efficacy of heterologous boosting against SARS-CoV-2 using a recombinant interferon-armed fusion protein vaccine (V-01): a randomized, double-blind and placebo-controlled phase III trial. Emerg Microbes Infect. 2022 Dec;11(1):1910-1919. doi: 10.1080/22221751.2022.2088406. PMID 35686572